| BioLite, Inc. | Protocol No.: BLI-1008-001 | Confidential |
|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

NCT Number: NCT0269908



# Statistical Analysis Plan (SAP)

# A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in Adult Patients with Attention-Deficit Hyperactivity Disorder (ADHD), Part I

PROTOCOL NUMBER BLI-1008-001

STUDY MEDICATION PDC-1421 Capsule

**SPONSOR** BioLite, Inc.

2F, No. 20, Sec. 2, Shengyi Rd., Zhubei City,

Hsinchu County 30261, Taiwan

**DATE** 17 Aug. 2020

VERSION 2.0

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

## **Comparison Table of SAP**

Original version: 1.0; Date: 2020/05/07. Revised version: 2.0; Date: 2020/08/17.

| Page 9 Protocol Number Page 14 3. Study Design Page 16 6.2 Treatment Sehedule Page 18-19 7. Protocol Versions and Protocol Amendments Page 18-19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) Page 20 Statistical Analysis Plan, Version: 2.0 Statisti | Changed items and | Version 1.0 | Version 2.0 | |
|---|---|---|---|---|
| All pages version Statistical Analysis Plan, Version: 2.0 BLI-1008- 001_protocol_v1.9_2020/01/15 Date: 7 May 2020 Page 9 BLI-1008-001 (Version 1.9) Protocol Number Page 14 3. Study Design Part I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30" Add the summary of statistical changes for protocol Amendments Page 19 (None) Add the statement "Round down to an integer." Add the statement "Round down to an integer." Add the statement is deleted. Page 20 Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health Page 10-108-001 (Version 2.0 Due to the sponsor's decision | | | AND THE RESERVE OF THE PARTY OF | Reasons |
| Version: 1.0 BLI-1008- 001_protocol_v1.9_2020/01/15 Date: 7 May 2020 Page 9 BLI-1008-001 (Version 1.9) Protocol Number Page 14 3. Study Design Part I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol Version 2.0. Page 19 (None) Add the summary of statistical changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Add the statement "Round down to an integer." Low to the sponsor's decision The targeted population of this Part I study is six subjects who met the per-protocol Agenta. Page 18-19 (None) Add the statement "Buring the CoVID-19 public health emergency, the assessments of CAARS or a mination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Low to the sponsor's decision The statement is deleted. Due to the sponsor's decision | | | | |
| BLI-1008- 001_protocol_v1.9_2020/01/15 Date: 7 May 2020 Page 9 Protocol Number Page 14 3. Study Design The targeted population of this Part I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule (None) (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) The T-scores of the subscales will be online calculated by a tool from Multi-Health The targeted population of this Part I study is six subjects who met the-per-protocol fine the targeted population of this Part I study is six subjects who met the-per-protocol fine the table, and the table protocol fine the table part I study is six subjects who met the-per-protocol fine the table, and the table part I study is six subjects who met the-per-protocol fine the table, and the table part I study is six subjects who met the-per-protocol fine the table, and the table part I study is six subjects who met the-per-protocol fine the table, and the satement "Ouring the definition more clearly The statement is deleted. Due to the sponsor's decision | All pages version | | | Version changed |
| Date: 7 May 2020 Page 9 Protocol Number Page 14 The targeted population of this part I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule (None) (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, CSSRS, AE evaluation, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18–19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) (None) (None) Add the statement "Round down to an integer." The targeted population of this Part I study is six subjects who met the per-protocol lassis. Page 18-19 CAARS, CGI, ADHDRS, CSSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the statement "Round definition more clearly Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health The targeted population of this Part I study is six subjects who met the-per-protocol (Version 2.0) Add the statement "Bound down to an integer." Due to protocol amendment definition more clearly Due to the sponsor's decision | | Version: 1.0 | Version: 2.0 | |
| Date: 7 May 2020 Page 9 Protocol Number Page 14 The targeted population of this part I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule (None) (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, CSSRS, AE evaluation, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18–19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) (None) (None) Add the statement "Round down to an integer." The targeted population of this Part I study is six subjects who met the per-protocol lassis. Page 18-19 CAARS, CGI, ADHDRS, CSSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the statement "Round definition more clearly Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health The targeted population of this Part I study is six subjects who met the-per-protocol (Version 2.0) Add the statement "Bound down to an integer." Due to protocol amendment definition more clearly Due to the sponsor's decision | | DI I 1000 | DI I 1000 | |
| Page 9 Protocol Number Page 14 Ref I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule Page 18 Ref I study is six subjects who met the per-protocol basis. Page 18 Ref I study is six subjects who met the per-protocol basis. Page 19 Ref I study is six subjects who met the per-protocol basis. Page 16 Ref I study is six subjects who met the per-protocol basis. Page 16 Ref I study is six subjects who met the per-protocol basis. Page 17 Ref I study is six subjects who met the per-protocol basis. Page 18 Ref I study is six subjects who met the per-protocol intent-to-treat basis. Page 19 Ref I study is six subjects who met the per-protocol intent-to-treat basis. Page 19 Ref Ref I study is six subjects who met the per-protocol intent-to-treat basis. Page 19 Ref Ref I study is six subjects who met the per-protocol intent-to-treat basis. Page 19 Ref Ref I study is six subjects who met the per-protocol intent-to-treat basis. Page 19 Ref | | | | |
| Page 9 Protocol Number Page 14 The targeted population of this 3. Study Design Part I study is six subjects who met the per-protocol basis. Page 16 (None) (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18–19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) BLI-1008-001 (Version 2.0) The targeted population of this Part I study is six subjects who met the per-protocol hais is subject who met the per-protocol intent-to-treat basis. Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) The T-scores of the subscales will be online calculated by a tool from Multi-Health The targeted population of this Part I study is six subjects who met the per-protocol intent-to-treat basis, and part I study is six subjects who met the per-protocol intent-to-treat basis. Part I study is six subjects who met the per-protocol intent-to-treat basis. Part I study is six subjects who met the per-protocol intent-to-treat basis. Add the statement "During the definition of the part of the per-protocol version 2.0" Add the statement "Round down to an integer." definition more clearly Due to the sponsor's decision | | 001_protocol_V1.9_2020/01/15 | 001_protocol_v2.0_2020/06/30 | |
| Page 9 Protocol Number Page 14 The targeted population of this 3. Study Design Part I study is six subjects who met the per-protocol basis. Page 16 (None) (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18–19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) BLI-1008-001 (Version 2.0) The targeted population of this Part I study is six subjects who met the per-protocol hais is subject who met the per-protocol intent-to-treat basis. Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) The T-scores of the subscales will be online calculated by a tool from Multi-Health The targeted population of this Part I study is six subjects who met the per-protocol intent-to-treat basis, and part I study is six subjects who met the per-protocol intent-to-treat basis. Part I study is six subjects who met the per-protocol intent-to-treat basis. Part I study is six subjects who met the per-protocol intent-to-treat basis. Add the statement "During the definition of the part of the per-protocol version 2.0" Add the statement "Round down to an integer." definition more clearly Due to the sponsor's decision | | Date: 7 May 2020 | Date: 17 Aug. 2020 | |
| Protocol Number Page 14 The targeted population of this 3. Study Design Part I study is six subjects who met the per-protocol basis. Page 16 (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18–19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) The targeted population of this Part I study is six subjects who met the per-protocol basis. Part I study is six subjects who met the per-protocol intent-to-treat basis. Part I study is six subjects who met the per-protocol treat basis. Add the statement "During the definition more clearly Page 18 Page 18 Page 18 Page 19 None) Add the statement "Round down to an integer." definition more clearly Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health | Page 9 | | _ | |
| 3. Study Design Part I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule Royard I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule Royard I study is six subjects who met the per-protocol intent-io-treat basis. Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18–19 7. Protocol Versions and Protocol Amendments Royard I study is six subjects who met the per-protocol intent-io-treat basis. Due to protocol amendment mendment of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) Royard Basis. Due to protocol amendment Specifying the definition more clearly The statement is deleted. Due to the sponsor's decision | Protocol Number | , | | |
| 3. Study Design Part I study is six subjects who met the per-protocol basis. Page 16 6.2 Treatment Schedule Roote I CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments Roote I Mone) Roote I Mone) Add "Version 2.0" and "2020/06/30". Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments Roote I Mone) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) The T-scores of the subscales will be online calculated by a tool from Multi-Health The statement is deleted. Due to the sporsor's decision | Page 14 | The targeted population of this | The targeted population of this | |
| Page 16 6.2 Treatment Schedule Region (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) (None) (None) Add the statement "Round down to an integer." The statement is deleted. Due to protocol amendment Due to protocol amendment Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) The T-scores of the subscales will be online calculated by a tool from Multi-Health | 3. Study Design | Part I study is six subjects who | Part I study is six subjects who | |
| Page 16 6.2 Treatment Schedule (None) Add the statement "During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments (None) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Due to protocol amendment Due to protocol amendment The statement is deleted. Due to the sponsor's decision Due to protocol amendment Due to protocol amendment The statement is deleted. Due to the sponsor's decision | | met the per-protocol basis. | met the per-protocol intent-to- | |
| COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments (None) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) (None) Add the statement "Round down to an integer." Jensel 19 Add the statement is deleted. The statement is deleted. Due to protocol amendment amendment amendment amendment by the protocol version 2.0. The statement is deleted. Due to the sponsor's decision | | | trcat basis. | |
| emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) (None) (None) Add the statement "Round down to an integer." Add the statement "Round definition more clearly The statement is deleted. Due to protocol amendment Due to protocol amendment Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) The statement is deleted. Due to the sponsor's decision | Page 16 | (None) | Add the statement "During the | |
| CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) (None) Add the statement "Round down to an integer." The statement is deleted. Due to protocol amendment Due to protocol amendment Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Specifying the definition more clearly The statement is deleted. Due to the sponsor's decision | 6.2 Treatment Schedule | | COVID-19 public health | |
| SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 (None) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) (None) Add the statement "Round down to an integer." Add the specifying the definition more clearly Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health Due to the sponsor's decision | | | emergency, the assessments of | |
| Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Page 18–19 7. Protocol Versions and Protocol Amendments (None) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 9.1 Age (years) (None) Add the statement "Round down to an integer." The T-scores of the subscales will be online calculated by a tool from Multi-Health Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Specifying the definition more clearly Due to the spoisor's decision | | | CAARS, CGI, ADHDRS, C- | |
| Page 18~19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) The <i>T</i> -scores of the subscales will be online calculated by a tool from Multi-Health Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Specifying the definition more clearly The statement is deleted. Due to the sponsor's decision | | | SSRS, AE evaluation, | Due to protocol |
| conducted by telephone, video, or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) (None) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Add the statement "Round down to an integer." definition more clearly The T-scores of the subscales will be online calculated by a tool from Multi-Health | | | Concomitant Medication, | amendment |
| or email, but those remote assessments should be documented." Page 18~19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) The T-scores of the subscales 9.5 CAARS-S:S will be online calculated by a tool from Multi-Health One of email, but those remote assessments should be documented." Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Specifying the definition more clearly The statement is deleted. Due to the sponsor's decision | | | Physical examination can be | |
| Page 18~19 (None) Page 18~19 (None) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Page 20 Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health assessments should be documented." Add theversion 2.0" and "2020/06/30". Add the statement "Round definition more clearly The statement is deleted. Due to the sponsor's decision | | | | |
| Page 18~19 (None) Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health Commonwealth | | | or email, but those remote | |
| Page 18~19 7. Protocol Versions and Protocol Amendments Page 19 9.1 Age (years) The <i>T</i> -scores of the subscales will be online calculated by a tool from Multi-Health Add "Version 2.0" and "2020/06/30". Add the summary of statistical changes for protocol version 2.0. Specifying the definition more clearly The statement is deleted. Due to the sponsor's decision | | | | |
| 7. Protocol Versions and Protocol Amendments Add the summary of statistical changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Page 20 Page 20 The <i>T</i> -scores of the subscales will be online calculated by a tool from Multi-Health "2020/06/30". Add the summary of statistical changes for protocol version 2.0. The statement "Round definition more clearly The statement is deleted. Due to the sponsor's decision | | | documented." | |
| Protocol Amendments Add the summary of statistical changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Page 20 Page 20 The <i>T</i> -scores of the subscales will be online calculated by a tool from Multi-Health Add the summary of statistical changes for protocol version 2.0. The statement "Round definition more clearly The statement is deleted. Due to the sponsor's decision | | (None) | | |
| changes for protocol version 2.0. Page 19 (None) Add the statement "Round down to an integer." Page 20 Page 20 The <i>T</i> -scores of the subscales 9.5 CAARS-S:S will be online calculated by a tool from Multi-Health | | | | |
| Page 19 (None) Add the statement "Round down to an integer." Page 20 Page 20 The <i>T</i> -scores of the subscales will be online calculated by a tool from Multi-Health 2.0. The statement "Round definition more clearly The statement is deleted. Due to the sponsor's decision | Protocol Amendments | | 1 | |
| Page 19 (None) Add the statement "Round down to an integer." Specifying the definition more clearly Page 20 The T-scores of the subscales will be online calculated by a tool from Multi-Health Add the statement "Round down to an integer." The statement is deleted. Due to the sponsor's decision | | | | |
| 9.1 Age (years) Page 20 Page 20 The <i>T</i> -scores of the subscales 9.5 CAARS-S:S will be online calculated by a tool from Multi-Health definition more clearly The statement is deleted. Due to the sponsor's decision | Page 10 | (None) | | Smooifring the |
| Page 20 The <i>T</i> -scores of the subscales 9.5 CAARS-S:S will be online calculated by a tool from Multi-Health clearly | | (None) | | |
| Page 20 The <i>T</i> -scores of the subscales will be online calculated by a tool from Multi-Health The statement is deleted. Due to the sponsor's decision | 9.1 Age (years) | | down to an integer. | |
| 9.5 CAARS-S:S will be online calculated by a tool from Multi-Health decision | Page 20 | The T-scores of the subscales | The statement is deleted | - |
| tool from Multi-Health | | | The Statement is defeted. | 1 |
| | 7.0 C. II II O D. O | | | |
| Systems Inc. Unline | | Systems Inc. Online | | |
| Assessment Center <sup>+</sup> . | | | | |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

| Changed items and | Version 1.0 | Version 2.0 | D |
|---|---|---|---|
| pages (new version) | Date: 2020/05/07 | Date: 2020/08/17 | Reasons |
| Page 25 | The <i>T</i> -scores of CAARS-S:S | The <i>T</i> -scores of CAARS-S:S | |
| 10.7.2 Secondary | will be assessed for each visit | (Conners et al. 1999) will be | |
| Efficacy Analyses | change from baseline (V3-V2, | assessed for each visit change | |
| | V4-V2,···,V8-V2) by | from baseline (V3-V2, V4- | |
| | Wilcoxon signed-rank test. | V2,···,V8-V2) by Wilcoxon | |
| | | signed-rank test. | Specifying the |
| Page 28 | (None) | Add the reference "Conners, C. | reference of T- |
| 12. Reference | | K., Erhardt, D., & Sparrow, E. | scores' calculation |
| | | P. (1999). Conners' adult | |
| | | ADHD rating scales (CAARS): | |
| | | technical manual. North | |
| | | Tonawanda, NY: Multi-Health | |
| | | Systems." | |
| Table T09.2~T09.3 | (None) | Indent the sub-items of | Being easier to read |
| | | "Relation to Study Drug" | |
| Listing | Listing L01.2: Listing of | The listing is deleted. | This should not be |
| | Protocol Deviation / Violation | | stated in SAP. |
| Listing | Listing L01.3 | Listing L01.2 | Recoding the |
| Listing | Listing L01.4 | Listing L01.3 | number |
| Listing L10.1~L10.2 | The content was presented as | The content is presented as | |
| | string. | number and the footnotes are | |
| | | added. | |
| Listing L11 | The content was presented as | The content is presented as | Due to the sponsor's |
| | string. | number and the footnotes are | decision |
| | | added. | |
| Listing L12.1~L12.3 | The content was presented as | The content is presented as | |
| | string. | number and the footnotes are | |
| | | added. | |
| Listing L13.1 | *(SAP, 9.6.3) | *The number of item is coded | Specifying the |
| | | in SAP, 9.6.3. | description more |
| | m | m | clearly |
| Listing L13.2 | The content was presented as | The content is presented as | Due to the sponsor's |
| | string. | number and the footnotes are | decision |
| Listing I 16 1-I 16 2 | (None) | added. Add the column "Series No." | Distinguishing the |
| Listing L16.1~L16.2 | (None) | | Distinguishing the data from different |
| Listing L17.1~L17.2 | (None) | Add the column "Series No." | time for each |
| | | | subject |
| | | | Subject |

| | 1 1000C01140 DL1-1000-001 | | Confidential |
|---|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 | CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

## Signature Page

SAP Author:

Wen-Jin Guo

Institute of Population

Health Sciences, National

Health Research Institutes

18/

Date

(DD/MMM/YYYY)

SAP Reviewer:

Chin-Fu Hsiao

Deputy Director,

Institute of Population

Health Sciences, National

Health Research Institutes

Signature

Date

(DD/MMM/YYYY)

Sponsor:

Chi-Hsin R. King

CSO,

New Drug Development

Division, BioLite, Inc.

ure

Date

(DD/MMM/YYYY)

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

## **Abbreviations and Definitions of Terms**

| Abbreviation | Term |
|---|---|
| Abn. w S. | Abnormal with significance |
| Abn. w/o S. | Abnormal without significance |
| ADHD | Attention-Deficit/Hyperactivity Disorder |
| ADHD-RS-IV | Attention-Deficit/Hyperactivity Disorder Rating Scale-IV |
| ADL | Activities of Daily Living |
| AE | Adverse Event, whether or not considered related to the investigational |
| | drug, must be recorded in CRF. |
| ALT | Alanine transaminase |
| aPTT | Activated partial thromboplastin time |
| AST | Aspartate aminotransferase |
| BUN | Blood Urea Nitrogen |
| C# | Category # (e.g. 'C6' means 'Category 6') |
| C-SSRS | Columbia-Suicide Severity Rating Scale |
| CAARS-S:S | Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale- |
| | Self Report: Short Version |
| CGI-ADHD-I | Clinical Global Impression-Attention-Deficit/Hyperactivity Disorder- |
| | Improvement |
| CGI-ADHD-S | Clinical Global Impression-Attention-Deficit/Hyperactivity Disorder- |
| | Severity |
| Clinical monitor | The designated CRA monitoring this study for the sponsor |
| CRA | Clinical Research Associate |
| CRC | Clinical Research Coordinator |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| CTCAE | Common Terminology Criteria for Adverse Events |
| DBP | Diastolic Blood Pressure |
| DSM-V | The Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition |
| ECG | The Electrocardiogram (ECG) is a graphical recording of the cardiac |
| | cycle produced by an electrocardiograph. |
| HCG | Human chorionic gonadotropin |
| HDL | High-Density Lipoprotein |
| HIV | Human Immunodeficiency Virus |
| HPLC | High Performance Liquid Chromatography |
| ICH | International Council for Harmonisation of Technical Requirements for |
| | Pharmaceuticals for Human Use |
| INR | International normalized ratio |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

## **Abbreviations and Definitions of Terms**

| Abbreviation | Term |
|---|---|
| IR | Infrared |
| ITT | Intent-to-Treat |
| LDH | Lactate Dehydrogenase |
| LDL | Lower-Density Lipoprotein |
| NLT | Not Less Than |
| NMT | Not More Than |
| p.o. | By mouth or orally |
| PP | Per-protocol |
| P.R.N. | pro re nata, a Latin phrase meaning "as needed." |
| PT | Prothrombin time |
| QTc | Q-T Interval Corrected For Heart Rate |
| RBC | Red Blood Cell |
| SAE | Serious Adverse Event, whether or not considered as related to the |
| | investigational drug must be recorded and reported. |
| SAP | Statistical Analysis Plan |
| SBP | Systolic Blood Pressure |
| Study Cohort | The Study Cohort is defined as a group or cohort of subjects who are |
| | assigned to take the same dose level of the study drug. |
| SUSAR | Serious and Unexpected Suspected Adverse Reaction |
| TID | Three times a day |
| TLC | Thin Layer Chromatography |
| TSH | Thyroid-stimulating hormone |
| UV | Ultraviolet |
| V# | Visit # (e.g. 'V6' means 'Visit 6') |
| WBC | White Blood Cell |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

## **Table of Contents**

| Abl | Abbreviations and Definitions of Terms | |
|---|---|---|
| Tal | Table of Contents | |
| 1. | Protocol Summary9 | |
| 2. | Tria | l Objectives |
| | 2.1 | Primary Objective |
| | 2.2 | Secondary Objective |
| 3. | Stud | ly Design |
| 4. | Stud | ly Endpoints |
| | 4.1 | Primary Endpoint |
| | 4.2 | Secondary Endpoints |
| | 4.3 | Safety Evaluation |
| 5. | Ran | domization and Blinding |
| 6. | Trea | ttment of Subjects |
| | 6.1 | Description of Study Drug |
| | 6.2 | Treatment Schedule |
| | 6.3 | Other Medication During the Study |
| 7. | | ocol Versions and Protocol Amendments |
| 8. | | ing and Operating Procedures for Final Analysis |
| 9. | Defi | nitions |
| | 9.1 | Age (years) 19 |
| | 9.2 | Treatment Compliance (%) |
| | 9.3 | ADHD-RS-IV |
| | 9.4 | Clinical Global Impression |
| | 9.5 | CAARS-S:S |
| | 9.6 | C-SSRS |
| 10. | Stat | istical Methodology |
| | 10.1 | Analyzed Populations |
| | 10.2 | Sample Size Determination |
| | 10.3 | Data Handling |
| | 10.4 | General Statistical Methodology |
| | 10.5 | Disposition of Subjects |
| | 10.6 | Demographic and Baseline Characteristics |
| | 10.7 | Efficacy Analyses |
| | 10.8 | Safety Analyses |
| 11. | Prog | gramming Considerations |
| | 11.1 | Statistical Software and Format of Output |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

## **Table of Contents**

| | 11.2 SAS Procedures for Descriptive/Inferential Statistics | . 27 |
|-----|------------------------------------------------------------|------|
| 12. | Reference | |
| 13. | Appendix | . 28 |
| | 13.1 Normal Range of Laboratory Tests | . 28 |
| | 13.2 Mock-up Tables | . 28 |
| | 13.3 Mock-up Patient Data Listings | 28 |

|---|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 | CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

## 1. Protocol Summary

| Name of Sponsor | BioLite, Inc. |
|---|---|
| Name of Finished | PDC-1421 Capsule |
| Product | |
| Name of Active | Name of Active PDC-1421 |
| Ingredient | |
| Study Title | A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in |
| | Adult Patients with Attention-Deficit Hyperactivity Disorder (ADHD), |
| | Part I |
| Clinical Trial Phase | II |
| Protocol Number | BLI-1008-001 (Version 2.0) |
| Principal Investigator | Dr. Keith McBurnett |
| Study Site | University of California San Francisco (UCSF) Medical Center |
| Study Period | 1 year |
| Study Objectives: | |
| Primary Study | To determine the efficacy profile of PDC-1421 Capsule in ADHD with |
| Objective | ADHD Rating Scale-IV (ADHD-RS-IV). |
| Secondary Study To determine the efficacy and safety profile of PDC-1421 Capsulo | |
| Objective | ADHD with other rating scales. |
| Methodology: | |
| Study Design | Part I: open label, dose escalation study |
| Number of Subjects | Maximum 6 subjects |
| <b>Duration of treatment</b> | 56 days |
| Study Intervention | The screening phase is intended for diagnosing and assessing the patient |
| | for possible inclusion in the study and for providing an adequate |
| | washout period. |
| | Part I is an open-label study, single center and dose escalation evaluation |
| in six subjects. Six subjects will be initially evaluated for safety a | |
| | efficacy assessments at low-dose (1 capsules TID) for 28 days. A safety |
| | checkpoint will be evaluated at day-28 for entering the high-dose (2 |
| | capsules TID). The subjects who pass the checkpoint will be initially |
| | evaluated for safety and efficacy assessments at high-dose (2 capsules |
| | TID) for 28 days. There will be an evaluation with all safety assessments |
| | data to decide whether this study passes the checkpoint to enter Part II. |
| Diagnosis and Main Criteria: | |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

| Study Population | Patients with ADHD according to the Diagnosis and Statistical Manual |
|---|---|
| | of Mental Disorders, 5th Edition |
| Inclusion Criteria | 1. Aged 18-70 years |
| | <ol> <li>Female subjects of child-bearing potential must test negative to pregnancy and use appropriate birth control method from the beginning of study to the 15 days later after ending of study</li> <li>Subjects must be able to understand and willing to sign informed consent</li> <li>Able to discontinue the use of any psychotropic medications for the treatment of ADHD symptoms at screening</li> <li>Meet strict operational criteria for adult ADHD according to the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V)</li> </ol> |
| | <ul> <li>6. A total score of 20 or higher on the 12-item ADHD index of Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) at screening</li> <li>7. Have a moderate or severe symptom of ADHD with score of 4 or higher in Clinical Global Impression-ADHD-Severity (CGI-ADHD-S) at screening</li> </ul> |
| Exclusion Criteria | <ol> <li>Have any clinically significant concurrent medical condition (endocrine, renal, respiratory, cardiovascular, hematological, immunological, cerebrovascular, neurological, anorexia, obesity or malignancy) that has become unstable and may interfere with the interpretation of safety and efficacy evaluations</li> <li>Have any clinically significant abnormal laboratory, vital sign, physical examination, or electrocardiogram (ECG) findings at screening that, in the opinion of the investigator, may interfere with the interpretation of safety or efficacy evaluations</li> <li>Have known serological evidence of human immunodeficiency virus (HIV) antibody</li> <li>Are pregnant as confirmed by a positive pregnancy test at screening</li> <li>Have QTc values &gt;450 msec at screening using Fridericia's QTc formula</li> <li>Have current of bipolar and psychotic disorders</li> <li>Have a current major depression disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder, panic disorder and eating disorder (also if treated but not currently symptomatic)</li> <li>NOTE: Comorbid diagnoses identified during screening and baseline are acceptable provided that ADHD is the primary</li> </ol> |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

| | diagnosis and the comorbid diagnoses will not confound study data or impair subject's ability to participate (per the Investigator's judgement and documented in source note). 8. Have any history of a significant suicide attempt, or possess a current risk of attempting suicide, in the investigator's opinion, based on clinical interview and responses provided on the Columbia-Suicide Severity Rating Scale (C-SSRS). 9. Have a history of jailing or imprisonment in the past 6 months due to worsening of symptoms of ADHD. |
|---|---|
| Early Withdrawal of | Subjects will be withdrawn from this trial if they meet one of the |
| Subjects | following withdrawal criteria: |
| | Subjects wish to withdraw. (Subjects are not obligated to give |
| | reasons for discontinuation from this trial.) |
| | Subjects can't obey the regulation of the study. |
| | • Investigator considers that withdrawal from study is the best interest |
| | of a subject. |
| | • The subject is pregnant during the trial. |
| | Subjects withdrawn from the study due to adverse event(s) must be |
| | followed until the events are recovered, recovered with residual effects, |
| Premature | death, or lost to follow-up. The Investigator and/or the Sponsor may decide to stop the trial if: |
| Termination or | Safety assessment clearly indicates that one study arm is associated |
| Suspension of the | with more severe or serious adverse experiences. |
| Study | The Sponsor decides to terminate the trial if necessary. |
| Test Product, Dose and | Regimen: |
| Name | PDC-1421 Capsule |
| Ingredients | PDC-1421: 380 mg, Silicon dioxide: 10 mg, Magnesium stearate: 10 |
| | mg. |
| Physical Appearance | Yellowish Granules in brownish capsule. |
| Loss on Drying | NMT 6% |
| Water Extractives | NLT 80% |
| Dilute-Alcohol | NLT 70% |
| Extractives | |
| Total Ash | NMT 5% |
| Acid-Insoluble Ash | NMT 4% |
| Alcohol Extractives | NLT 38% |
| TLC | 1. One grayish blue band has same $R_f$ value as reference standard (3',6- |
| | disinapoylsucrose); |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

| | 2. One watchet blue band has same R <sub>f</sub> value as reference standard |
|---|---|
| | (Glomeratose A). |
| HPLC of Markers | 1. $10.0 \text{ mg/g} \le \text{Glomeratose A} \le 30.0 \text{ mg/g}$ . |
| | 2. 38 mg/g ≤ 3',6-Disinapoylsucrose ≤ 95 mg/g. |
| UV Spectrum | λ <sub>max</sub> : 230~240 nm; 315~325 nm |
| IR Spectrum (cm <sup>-1</sup> , | Peak at: $3380 \pm 100$ Broad, $2938 \pm 20$ Sharp, $1605 \pm 10$ Sharp, $1455 \pm$ |
| <b>%T</b> ) | 10 Sharp, $833 \pm 10$ Sharp. |
| pН | Dissolved in distill deionized water at a concentration of 0.1 g/ml, $3.8 \le$ |
| | pH ≤5.8. |
| Uniformity | 90~110% |
| Weight Variation | 90~110% |
| Heavy Metal | Cu < 20 ppm, As < 1 ppm, Pb < 5 ppm, Cd < 0.2 ppm, Hg < 0.1 ppm |
| | Total aerobic plate count: NMT 10 <sup>3</sup> CFU/g |
| | Mold and yeast count: NMT 100 CFU/g |
| Microbial Purity | Echerichia coli: Undetectable |
| | Staphylococcus aureus: Undetectable |
| | Salmonella: Undetectable |
| Dose and Regimen | 1 and 2 capsules thrice daily, p.o., after meal |
| Clinical Endpoints: | |
| Primary Endpoint | Improvement of 40% or greater in ADHD Rating Scale-Investigator |
| | Rated (ADHD-RS-IV) from baseline up to 8 weeks treatment |
| Secondary Endpoints | Change from baseline in the Conners' Adult Attention- |
| | Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short |
| | Version (CAARS-S:S) to 8 weeks treatment. |
| | Clinical Global Impression-ADHD-Severity (CGI-ADHD-S) and |
| | Clinical Global Impression-ADHD-improvement (CGI-ADHD-I) |
| | score of 2 or lower. |
| Safety Evaluation | A. Change from baseline in: |
| | 1. vital sign |
| | 2. physical examination |
| | 3. electrocardiogram (ECG) |
| | 4. laboratory tests (hematology and biochemistry) |
| | B. Incidence of AE/SAE |
| | C. Suicidal ideation and behavior by Columbia-Suicide Severity Rating |
| | Scale (C-SSRS) |
| Statistical Consideratio | ns: |
| Statistical Consideration Sample Size | In part I study, six subjects each will be evaluated for safety and efficacy |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | 5 Date: 17 Aug. 2020 |

| Determination | assessments at 1 and then 2 capsules TID dose for total 56 days (28 days |
|---|---|
| | at each dose). |
| General Statistical | 1. Subjects Population |
| Methodology | <ul> <li>Intent-to-Treat (ITT) Population: The data are analyzed on patients who take at least one dose of study medication and have any post-baseline measurements collected.</li> <li>Per-protocol (PP) Population: <ul> <li>The drug compliance is at least 80%</li> <li>Subjects have completed data to determine the primary endpoint.</li> <li>Subjects cannot have protocol deviation.</li> <li>Safety Population: The safety measures are conducted on the patients who take at least one dose of study medication.</li> </ul> </li> <li>Statistical Method <ul> <li>Simple descriptive statistics with 95% confidence interval will be performed with data collected in this study wherever applicable. All data shall be tabulated and presented in the study report. The safety and efficacy data will be analyzed using the non-parametric method wherever appropriate.</li> </ul> </li> </ul> |
| | The purpose for Part I is exploratory in safety and the formal statistical analysis will not be needed. The descriptive statistics will be provided. Safety endpoints will be listed and summarized as |
| | appropriate: median and range for continuous data; frequencies, total numbers and percentages for categorical data. |

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

#### 2. Trial Objectives

#### 2.1 Primary Objective

The objective of this trial was to determine the effective doses and treatment period of PDC-1421 Capsule in subjects with ADHD.

#### 2.2 Secondary Objective

The objective was to evaluate the safety of PDC-1421 Capsule in subjects receiving PDC-1421 at various dose levels.

#### 3. Study Design

The Screening phase is intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. The targeted population of this Part I study is six subjects who met the intent-to-treat basis. Part I study is an open-label study, single center and dose escalation evaluation in six patients.



<u>Low dose</u>: Six subjects will be initially evaluated for safety and efficacy assessments at low-dose (1 capsule TID) for 28 days. Subject will return for visit once a week during treatment period.

<u>Checkpoint #1</u>: There will be an evaluation with all safety assessments data to decide whether you pass the checkpoint to enter high-dose treatment or continue to receive a low-dose treatment by the investigator.

<u>High dose</u>: The subjects who pass the checkpoint #1 will be initially evaluated for safety and efficacy assessments at high-dose (2 capsules TID) for 28 days. Subject will return for visit biweekly during treatment period.

<u>Checkpoint #2</u>: There will be an evaluation with all safety assessments data to decide whether this study passes the checkpoint to enter Part II by the investigators.

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

#### 4. Study Endpoints

4.1 Primary Endpoint

Improvement of 40% or greater in ADHD Rating Scale-Investigator Rated (ADHD-RS-IV) from baseline up to 8 weeks treatment.

- 4.2 Secondary Endpoints
  - 4.2.1 Change from baseline in the Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (CAARS-S:S) up to 8 weeks treatment.
  - 4.2.2 Clinical Global Impression-ADHD-Severity (CGI-ADHD-S) and Clinical Global Impression-ADHD-Improvement (CGI-ADHD-I) score of 2 or lower.
- 4.3 Safety Evaluation
  - 4.3.1 Change from baseline in:
    - vital sign
    - · physical examination
    - electrocardiogram (ECG)
    - laboratory tests (hematology and biochemistry)
  - 4.3.2 Incidence of AE/SAE
  - 4.3.3 Suicidal ideation and behavior by Columbia-Suicide Severity Rating Scale (C-SSRS)

#### 5. Randomization and Blinding

| | Part I |
|---------------|-------------------|
| Randomization | None (open label) |
| Blinding | None (open label) |

#### 6. Treatment of Subjects

6.1 Description of Study Drug

PDC-1421 Capsule is a botanical investigational new drug. Each PDC-1421 Capsule contains 380 mg PDC-1421 drug substance extracted from dry root of *P. tenuifolia*.

6.2 Treatment Schedule

Potential subjects will be introduced by Investigator of the study design at Screening. If the subject agrees to participate and signs the consent form, the screening process will begin. Suitability of the subject will be evaluated by inclusion/exclusion criteria.

In part I Study, six eligible subjects will receive a low-dose treatment with 1 PDC-1421 Capsule thrice daily for 28 days (4 weeks) and be assessed once a week (Visit 2, 3, 4, 5, and 6). After passing a dose-up checkpoint for the safety of individual subjects, these subjects will then receive a high-dose treatment with 2 PDC-1421 Capsules thrice daily for another 28 days (4 weeks). Subjects will be assessed every two weeks (Visit 6, 7 and 8) in high-dose treatment. After the end of part I Study, subjects will be requested to return for a follow-up visit (Visit 9) two weeks later after the last dose.

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

During the COVID-19 public health emergency, the assessments of CAARS, CGI, ADHDRS, C-SSRS, AE evaluation, Concomitant Medication, Physical examination can be conducted by telephone, video, or email, but those remote assessments should be documented.

| Procedure table: BLI-1008-001 protocol | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| *Week | -2 | 0 | 1 | 2 | 3 | 4 | 6 | 8 | 10 |
| Visit | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| DSM-V | $\checkmark$ | | | | | | | | |
| CAARS-S:S | √ | √ | √ | 1 | √ | $\sqrt{}$ | √ | √ | |
| CGI-ADHD-S | | √ | √ | 1 | √ | $\sqrt{}$ | √ | | |
| CGI-ADHD-I | | √ | √ | 1 | √ | $\sqrt{}$ | √ | | |
| ADHD-RS-IV | | √ | √ | √ | √ | $\sqrt{}$ | √ | | |
| C-SSRS | √ | √ | √ | 1 | √ | | √ | √ | √ |
| AE/SAE evaluation | | | √ | 1 | √ | √ | √ | √ | √ |
| Concomitant | | √ | √ | √ | | | √ | √ | |
| Medication | <b>'</b> | , v | <b>'</b> | , v | <b>'</b> | <b>'</b> | <b>'</b> | , v | |
| Physical | | | | | | | | √ | |
| examination | | | | | | | | | |
| Vital sign | √ | √ | √ | √ | √ | √ | √ | √ | |
| ECG | √ | | | | | | | √ | |
| Hematology | √ | √ | | 1 | | √ | √ | √ | |
| <b>Blood Chemistry</b> | √ | √ | | 1 | | √ | √ | √ | |
| Blood drawing | | V | | <b>√</b> | | V | | | |
| (venipuncture) | , v | \ \ \ | | , v | | , v | , v | , v | |
| Pregnancy test | √ | | | | | | | | √ |

<sup>\*</sup>On  $\pm 2$  days.

#### 6.2.1 Screening Phase (Visit 1)

The Screening phase will be done within 1~2 weeks period and intended for diagnosing and assessing the patient for possible inclusion in the study and for providing an adequate washout period. The items of physical, rating scales and laboratory examination at screening are outlined below:

- Informed consent
- Subject information, including date of birth, gender, body height and weight
- Medical history (within six month), including any clinically significant psychiatric, neurological, gastrointestinal, renal, hepatic, cardiovascular, respiratory, metabolic, endocrine, hematological or other major disorders
- Pregnancy test
- Physical examination: skin, head, neck, eyes, ears, nose, throat, heart, lungs, abdomen (liver, spleen), neurological examination, lymph node and extremities.

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

- Vital sign: heart rate, blood pressure, body temperature
- ECG
- Hematology: RBC, WBC, platelets, hematocrit, hemoglobin, prothrombin time (PT), partial thromboplastin time (aPTT)
- Blood chemistry: AST, ALT, LDH, total bilirubin, BUN, serum creatinine, free thyroxine (FT4), TSH, sodium, calcium, potassium, HbA1c, LDL, HDL, triglyceride, cholesterol
- DSM-V, CAARS-S:S, CGI-ADHD-S, ADHD-RS-IV, C-SSRS
- Concomitant medication evaluation
- Eligibility evaluation: laboratory data, other tests and evaluation results shall be obtained at Screening to determine the appropriateness of subject enrolled in this study

## 6.2.2 Part I Study. - Treatment Period (Visit 2~8) and Follow-up (Visit 9)

Subjects who meet the eligibility criteria will be enrolled and take test drug at this period. Six eligible subjects will take 1 capsule of PDC-1421 Capsule thrice daily for four weeks. They will receive a drug bag and be instructed to take 1 PDC-1421 Capsule thrice daily after meals. Weekly visits (Visit 2, 3, 4 and 5) will be requested during this 28-day treatment period. At Visit 6, all subjects will be evaluated with safety assessments and to be decided whether they will enter the high-dose treatment by the investigator. In the high-dose treatment, subjects will receive a drug bag and be instructed to take 2 PDC-1421 Capsule thrice daily after meals for 4 weeks. Biweekly visits (Visit 6, 7 and 8) will be requested during this 28-day treatment period. After two weeks of the last dose administration, subjects are assessed for a follow-up. Then, a checkpoint will be conducted. If subjects have no drug-related SAE, the schedule can be conducted to the part II. The items of safety and efficacy parameters at treatment period are outlined below:

- Physical examination: skin, head, neck, eyes, ears, nose, throat, heart, lungs, abdomen (liver, spleen), neurological examination, lymph node and extremities (only at Visit 8).
- Vital sign: heart rate, blood pressure, body temperature
- ECG (Only at Visit 8).
- Hematology: RBC, WBC, platelets, hematocrit, hemoglobin, prothrombin time (PT), partial thromboplastin time (aPTT) (Only at Visit 2,4,6,7 and 8).
- Blood chemistry: AST, ALT, LDH, total bilirubin, BUN, serum creatinine, free thyroxine (FT4), TSH, sodium, calcium, potassium, LDL, HDL, triglyceride, cholesterol (Only at Visit 2,4,6,7, and 8).
- CAARS-S:S, CGI-ADHD-S, CGI-ADHD-I, ADHD-RS-IV, C-SSRS and concomitant medication evaluation.
- AE/SAE evaluation (Subjects will not need to be assessed for AE/SAE at visit 2.)
- Drug accountability

| BioLit | e, Inc. | Protocol No.: BLI-1008-001 | | Confidential |
|---|---|---|---|---|
| Statisti | ical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 | CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

Follow-up visit will be performed at visit 9 after two weeks of the last dose administration. The test items are outlined in the following:

- C-SSRS.
- AE/SAE evaluation
- Pregnancy test

#### 6.3 Other Medication During the Study

To avoid conflict or unknown effects with the study drug, subjects are prohibited from taking any anti-ADHD medication and psychoactive drugs, as per the exclusion criteria, including MAOIs (monoamine oxidase inhibitor), NRIs (norepinephrine reuptake inhibitor) and norepinephrine receptor agonist/antagonist. Subjects can't combine the newly-initiated psychotherapy. If subjects have severe insomnia and are currently taking Zolpidem, Zopiclone or Zaleplon (sedative-hypnotics), they will be queried whether they can comply with the discontinuation:

- Subjects who indicate that they can discontinue will be washed out for 1 week, and then allowed to begin study protocol;
- Subjects who indicate that they are unable to discontinue will be allowed to enroll if they
  are able to agree that their use will be consistent and will not change for the duration of
  the study. (The maximum daily dose in Zolpidem, Zopiclone and Zaleplon are 10 mg,
  7.5 mg and 10 mg respectively.)

#### 7. Protocol Versions and Protocol Amendments

Approved versions of study protocol are listed as following.

| Version No. | Version Date |
|-------------|--------------|
| Version 1.2 | 2018/06/06 |
| Version 1.6 | 2019/03/22 |
| Version 1.7 | 2019/05/03 |
| Version 1.8 | 2019/07/26 |
| Version 1.9 | 2020/01/15 |
| Version 2.0 | 2020/06/30 |

Amendments relevant to statistical parts from version 1.2 to 2.0 are highlighted / crossed-out in table below:

#### Summary of statistical changes for protocol version 1.6

#### 8.3 Analysis of Efficacy and Safety

The statement "The comparison between three groups will be analyzed by nonparametric method as appropriate" was revised to "The comparison between two groups will be analyzed by nonparametric method as appropriate".

#### Summary of statistical changes for protocol version 1.7

No amendments on statistical parts.

## Summary of statistical changes for protocol version 1.8

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

No amendments on statistical parts.

#### Summary of statistical changes for protocol version 1.9

#### 8.2 Statistical Method

The first paragraph was revised to "Simple descriptive statistics with 95% confidence interval will be performed with data collected in this study wherever applicable. All data shall be tabulated and presented in the study report. The safety and efficacy data will be analyzed using the non-parametric method wherever appropriate."

- 8.3 Analysis of Efficacy and Safety
- The third item of definition of protocol deviation was deleted.
- The definition of an intent-to-treat (ITT) basis was revised to "the data are analyzed on patients who take at least one dose of study medication and have any post-baseline measurements collected."
- The statement "The safety measures are conducted on the ITT basis" was revised to "The safety measures are conducted on the patients who take at least one dose of study medication."
- The statement "The comparison between two groups will be analyzed by nonparametric method as appropriate" was deleted.

## Summary of statistical changes for protocol version 2.0

#### 3.1 General Design

The statement "The targeted population of this Part I study is six subjects who met the perprotocol basis" was revised to "The targeted population of this Part I study is six subjects who met the intent-to-treat basis."

#### 8. Timing and Operating Procedures for Final Analysis

The final analysis will be planned according to the study protocol. The timing of analysis and data to be cleaned is detailed as following:

- (1) Data to be cleaned: When 6 subjects have been recruited and all subjects are off study. All clinical trial data will be cleaned up for the analyses.
- (2) Timing of analysis: After all clinical trial data were cleaned up and the database will be locked for the final analysis. Then, all data will be analyzed according to SAP. Statistical programs will be prepared and executed by NHRI.

#### 9. Definitions

9.1 Age (years)

(Date of informed consent form signed–Date of Birth+1) / 365.25. Round down to an integer.

9.2 Treatment Compliance (%)

Subjects' compliance during the treatment period will be calculated according to the following formula:

Number of study medication actually took during the extent of exposure

Number of study medication should be taken during the extent of exposure (#)

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

# = (Number of study medication should be taken per day) \* (Extent of exposure).

Number of study medication actually took = quantity of dispensed capsules – quantity of returned capsules – quantity of lost capsules.

• Extent of exposure (days):

Extent of exposure before Checkpoint 1 = date of V6 - date of the first drug taken.

Extent of exposure after Checkpoint 1 = date of the last drug taken - date of V6 + 1.

Subjects' mean daily dose of the test drug will be calculated by

## Number of study medication actually took

#### Extent of exposure

- If the date of the first drug taken is not available, the date when the drug was firstly dispensed will be used for calculation.
- If the date of last drug taken is not available, the date will be replaced with that of the last drug return, previous drug taken, or previous drug return in order.

#### 9.3 ADHD-RS-IV

The ADHD-RS-IV with Adult Prompts is an 18-item scale base on the DSM-IV-TR' criteria for ADHD that provides a rating of the severity of symptoms. The adult prompts serve a guide to explore more fully the extent and severity of ADHD symptoms and create a framework to ascertain impairment. The odd-numbered 9 items assess inattentive symptoms and the even-numbered 9 items assess hyperactive-impulsive symptoms. Scoring is based on a 4-point, yielding a possible total score of  $0\sim54$ . Likert-type severity scale: 0 = Never or Rarely, 1 = Sometimes, 2 = Often, 3 = Very Often. Clinicians should score the highest score that is generated for the prompts for each item.

For inattention (IA) subscale raw score: Add the odd-numbered 9 items

For hyperactivity-impulsivity (HI) subscale raw score: Add the even-numbered 9 items To obtain the total raw score: Add the IA and HI subscale raw scores.

## 9.4 Clinical Global Impression

At the baseline visit, clinicians completed the CGI-S and were asked to evaluate the severity of subjects' illness with respect to ADHD symptoms based on the clinician's experience with this particular population. Possible scores ranged from 1 (normal, not ill at all) to 7 (among the most extremely ill subjects). At all subsequent study visits, clinicians used the CGI-I to rate the subjects' total improvement based on comparison with their baseline assessment from 1 (very much improved) to 7 (very much worse).

#### 9.5 CAARS-S:S

Conners' Adult Attention-Deficit/Hyperactivity Disorder Rating Scale-Self Report: Short Version (Conners et al., 1998; CAARS-S:S) consists of 26 items rated from 0 'not at all, never' to 3 'very much, very frequently.' Four subscales each composed of 5 items (A: Inattention/Memory Problems; B: Hyperactivity/Restlessness; C: Impulsivity/Emctional Lability; and D: Problems with Self-Concept) as well as a 12-item ADHD index can be computed. The CAARS-S:S was administered by computer-assisted personal interview (CAPI) prior to the first treatment session.

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

#### 9.6 C-SSRS

#### 9.6.1 Suicidal Ideation

The five boxes in the Suicidal Ideation, from the left to the right, of the CRF represents the five binary responses (yes/no) of the five items are as following.

- 1. Wish to be Dead (C1)
- 2. Non-Specific Active Suicidal Thoughts (C2)
- 3. Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act (C3)
- 4. Active Suicidal Ideation with Some Intent to Act, without Specific Plan (C4)
- 5. Active Suicidal Ideation with Specific Plan and Intent (C5)

#### 9.6.2 Intensity of Ideation

The first box of the six boxes in the Intensity of Ideation of the CRF records the most severe type of suicidal ideation. The remaining boxes, from the left to the right, represent the following items.

#### #1. Frequency

(1 = Less than once a week, 2 = Once a week, 3 = 2-5 times in week, 4 = Daily or almost daily, 5 = Many times each day)

#### #2. Duration

(1 = Fleeting – few seconds or minutes, 2 = Less than 1 hour/some of the time, 3 = 1-4 hours/a lot of time, 4 = 4-8 hours/most of day, 5 = More than 8 hours/persistent or continuous)

#### #3. Controllability

(1 = Easily able to control thoughts, 2 = Can control thoughts with little difficulty, 3 = Can control thoughts with some difficulty, 4 = Can control thoughts with a lot of difficulty, 5 = Unable to control thoughts, 0 = Does not attempt to control thoughts)

#### #4. Deterrents

(1 = Deterrents definitely stopped you from attempting suicide, 2 = Deterrents probably stopped you, 3 = Uncertain that deterrents stopped you, 4 = Deterrents most likely did not stop you, 5 = Deterrents definitely did not stop you, 0 = Does not apply)

#### #5. Reasons for Ideation

(1 = Completely to get attention, revenge or a reaction from others, 2 = Mostly to get attention, revenge or a reaction from others, 3 = Equally to get attention, revenge or a reaction from others and to end/stop the pain, 4 = Mostly to end or stop the pain, 5 = Completely to end or stop the pain, 0 = Does not apply)

#### 9.6.3 Suicidal Behavior

The boxes in the Suicidal Behavior, from the left to the right, of the CRF represents the binary responses (yes/no) of the items are as following.

- 6. Actual Attempt (C9)
- 7. Non-Suicidal Self-Injurious Behavior (Self-injurious behavior without suicidal

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

intent)

- 8. Interrupted Attempt (C8)
- 9. Aborted Attempt (C7)
- 10. Preparatory Acts or Behavior (C6)
- 11. Suicidal Behavior
- 12. Completed Suicide (C10, not available in screening)

#### 10. Statistical Methodology

#### 10.1 Analyzed Populations

#### 10.1.1 Intent-to-Treat (ITT) Population

The data are analyzed on patients who take at least one dose of study medication and have any post-baseline measurements collected.

#### 10.1.2 Per-protocol (PP) Population

- The drug compliance is at least 80%.
- Subjects have completed data to determine the primary endpoint.
- Subjects cannot have protocol deviation.

#### 10.1.3 Safety Population

The safety measures are conducted on the patients who take at least one dose of study medication.

#### 10.2 Sample Size Determination

In part I study, six subjects each will be evaluated for safety and efficacy assessments at 1 and then 2 capsules TID dose for total 56 days (28 days at each dose).

#### 10.3 Data Handling

#### 10.3.1 Definition of Baseline Values

The data obtained from eligible subjects before study drug administration in Visit 2 are set as baseline.

#### 10.3.2 Data Handling for Missing Data

The data are analyzed utilizing the last observation carried forward (LOCF) technique to impute the missing data.

#### 10.3.3 Definition of Protocol Deviation

- Inclusion or exclusion criteria not satisfied.
- · Not permitted concomitant medications.

#### 10.4 General Statistical Methodology

The purpose for Part I is exploratory in safety and the formal statistical analysis will not be needed. All data shall be tabulated and presented in the study report. The descriptive statistics will be provided. The efficacy and safety information recorded on CRF will be summarized by tables presented in frequency and percentage for categorical variables, in mean with SD as well as median with the minimum and maximum for continuous variables. All adverse events will be summarized with coding term, severity, relationship to study drug by frequency tables with the counts and percentage. In addition, serious adverse events will be

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

listed with event narration. Simple descriptive statistics with 95% confidence interval will be performed with data collected in this study wherever applicable. The safety and efficacy data will be analyzed using the non-parametric method wherever appropriate.

## 10.5 Disposition of Subjects

- Entered subject number
- Overall status and reason of withdraw / early termination

## 10.6 Demographic and Baseline Characteristics

#### 10.6.1 Demographic Characteristics

- Age
- Gender
- Height (cm)
- Weight (lb)

#### 10.6.2 Baseline Characteristics

- DSM-V (score)
  - Inattention Symptoms
  - Hyperactivity Symptoms
  - Impulsivity Symptoms
- ADHD-RS-IV (score)
  - Inattention Subscale
  - Hyperactivity-Impulsivity Subscale
  - Total Score
- CAARS-S:S (score)
  - Inattention/Memory Problems
  - Hyperactivity/Restlessness
  - Impulsivity/Emotional Lability
  - Problems with Self-Concept
  - ADHD index
- Clinical Global Impression (score)
  - Severity of illness
  - Improvement
- Physical Examinations
  - Skin
  - Head and Neck
  - Eyes
  - Ears
  - Nose
  - Throat
  - Heart
  - Lungs
  - Abdomen / liver, spleen

|---|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 | CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

- Extremities
- Neurological
- Lymph Node
- Vital Signs
  - Systolic Blood Pressure (mm/Hg)
  - Diastolic Blood Pressure (mm/Hg)
  - Heart Rate (bpm)
  - Temperature (°F)
- Electrocardiogram (ECG)
  - QTc value (msec)
- Hematology
  - RBC (g/dL)
  - WBC (x10<sup>3</sup>/mm<sup>3</sup>)
  - Hemoglobin (g/dL)
  - Hematocrit (%)
  - Platelet (x10<sup>3</sup>/mm<sup>3</sup>)
  - aPTT (sec)
  - PT (INR)
- Biochemistry
  - BUN (mg/dl)
  - Creatinine (mg/dl)
  - Total Bilirubin (mg/dl)
  - Sodium (mmol/L) (Na)
  - Calcium (mmol/L) (Ca)
  - Potassium (mmol/L) (K)
  - AST (U/L) (SGOT)
  - ALT (U/L) (SGPT)
  - LDH (U/L)
  - TSH (mui/ml)
  - Free T (ng/dl)
  - HbA1c (%)
  - LDL (mg/dL)
  - HDL (mg/dL)
  - Triglyceride (mg/dL)
  - Cholesterol (mg/dL)
  - HCG (Pregnancy Test)
- C-SSRS
  - Suicidal Ideation
  - Suicidal Behavior

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

#### 10.7 Efficacy Analyses

In part I study, efficacy assessments are conducted from screening stage to the last visit. Efficacy parameters are outlined as follows:

- ADHD-RS-IV
- Clinical Global Impression
- CAARS-S:S

#### 10.7.1 Primary Efficacy Analyses

- The scores of ADHD-RS-IV will be assessed by the descriptive statistics of tendency and variability.
- The improvement, which is greater than or equal to 40%, in ADHD-RS-IV from baseline up to 8 weeks (V3~V8) treatment will be summarized by way of frequency and percentage.

#### 10.7.2 Secondary Efficacy Analyses

- The *T*-scores of CAARS-S:S (Conners et al. 1999) will be assessed for each visit change from baseline (V3-V2, V4-V2,...,V8-V2) by Wilcoxon signed-rank test.
- The scores of 2 or lower of CGI-ADHD-S (V1~V8) and CGI-ADHD-I (V3~V8) will be summarized by way of frequency and percentage.

#### 10.8 Safety Analyses

Safety parameters are outlined as follows:

- Data collected from the physical examinations, vital sign, ECG and laboratory test in scheduled visit
- Adverse events reported
- Serious adverse events reported
- C-SSRS evaluation

The data obtained before study drug administration in Visit 2 are set as baseline. After the beginning of treatment, the collection of data of safety parameters are performed at planned treatment schedule as section 6.2. AE or SAE will be closely monitored during the study period. CRC shall record these data in CRF in detail. In part I, data are recorded from screening stage to the last visit.

#### 10.8.1 Adverse Event (AE)

Adverse event is any unfavorable and unintended symptom, syndrome, medical condition or experience that develops or worsens within the study period. In this Phase II trial, any clinically significant abnormal findings, including causing the subject to withdraw from the study, requiring treatment or causing apparent clinical manifestations, or judged relevant by the investigator, are considered to be AEs and will be monitored and recorded. AE may not be causal relationship with study medication or clinical study. Whether related to study medication or not, CRC shall record the information of AEs in CRF. The information of AEs contains characteristic, onset and duration, frequency, the Investigator's opinion of the relationship to the study drug (unrelated, unlikely, possibly, probably, definitely), outcome (recovered,

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

recovered with residual effects, continuing, death, lost to follow-up) and severity. Common Terminology Criteria for Adverse Events v4.03 (CTCAE) is a descriptive terminology and the grading (severity) scale is provided for each AE term. In the final analysis, all adverse events will be summarized with coding term, severity, relationship to study drug by frequency tables with the counts and percentage.

| Grade | Description |
|---|---|
| Grade 1 | Mild; asymptomatic or mild symptoms; clinical or diagnostic |
| | observations only; intervention not indicated. |
| Grade 2 | Moderate; minimal, local or noninvasive intervention indicated |
| | limiting age-appropriate instrumental activities of daily living (ADL)*. |
| Grade 3 | Severe or medically significant but not immediately life-threatening; |
| | hospitalization or prolongation of hospitalization indicated; disabling; |
| | limiting self-care ADL†. |
| Grade 4 | Life-threatening consequences; urgent intervention indicated. |
| Grade 5 | Death related to AE. |

<sup>\*</sup>Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

#### 10.8.2 Serious Adverse Event (SAE)

SAE is defined as any significantly untoward medical occurrence, including:

- Death
- Life-threatening condition
- Inpatient hospitalization or prolongation of existing hospitalization
- Persistent or significant disability/incapacity
- Congenital anomaly/birth defect
- Required intervention to prevent permanent impairment/damage

#### 10.8.3 Serious and Unexpected Suspected Adverse Reaction (SUSAR)

SUSAR is defined as any significantly untoward medical occurrence, the nature or severity of:

- Which is not consistent with the applicable product information (e.g., Investigator's Brochure) for an unapproved investigational medicinal product.
- Which must be causal relationship with study medication or clinical study.

#### 10.8.4 Other Safety Endpoints

- Physical examinations will be summarized for V8 change from V1 by way of frequency and percentage.
- Vital signs will be summarized for each treatment visit (V3~V8) change from baseline by way of frequency and percentage, and assessed by the descriptive statistics of tendency and variability.
- The ECG will be summarized for V8 change from V1 by way of frequency and percentage, and assessed by the descriptive statistics of tendency and variability.

<sup>†</sup>Self-care ADL refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

- Hematology will be summarized for some visits (V4, V6, V7, V8) change from baseline by way of frequency and percentage, and assessed by the descriptive statistics of tendency and variability.
- Biochemistry will be summarized for some visits (V4, V6, V7, V8) change from
  baseline by way of frequency and percentage except for HbA1c, and assessed by
  the descriptive statistics of tendency and variability. The HCG (pregnancy test)
  will be summarized for V9 change from V1 by way of frequency and percentage.
- C-SSRS (Nilsson et al. 2013)
  - Suicidal Ideation (C1~C5), Suicidal Behavior (C6~C10), and Self-Injurious Behavior without Suicidal Intent will be summarized for each visit (V1~V9) by way of frequency and percentage.
  - Some Suicide-Related Treatment-Emergent Events will be summarized by way of frequency and percentage.
  - Categories (C1~C10) will be summarized by a shift-table to demonstrate changes some visits (V3~V8) from baseline.
  - The most severe type of suicidal ideation will be summarized by a shift-table to demonstrate changes some visits (V3~V8) from baseline. We define no suicidal ideation as 0.

## 11. Programming Considerations

11.1 Statistical Software and Format of Output

Results presented in tables, figures and graphs (section 14 of ICH/CSR) and in patient data listing (section 16 of ICH/CSR) will be created with SAS version 9.4 or above. The format (mock-up table/figure and listing) can be found in Appendix.

11.2 SAS Procedures for Descriptive/Inferential Statistics

| Statistics | Relevant Syntax |
|----------------------------|-------------------------------------------------|
| Descriptive Statistics For | PROC FREQ |
| Categorical Variable | DATA = aaa; |
| Carregorieur variable | TABLES variable; |
| | RUN; |
| Descriptive Statistics For | PROC MEANS |
| Continuous Variable | DATA = bbb |
| Commuous variable | N MEAN STD MIN MEDIAN MAX LCLM UCLM ALPHA=0.05; |
| | VAR variable; |
| | RUN; |
| Wilcoxon signed-rank test | PROC UNIVARIATE |
| | DATA = ccc; |
| | VAR variable; |
| | RUN; |

#### 12. Reference

 A Phase II Tolerability and Efficacy Study of PDC-1421 Treatment in Adult Patients with Attention-Deficit Hyperactivity Disorder (ADHD), Part I (Protocol Number: BLI-1008-001)

|---|---|---|
| Statistical Analysis Plan, Version: 2.0 | BLI-1008-001_protocol_v2.0_2020/06/30 CRF Version 2.1_2020/03/16 | Date: 17 Aug. 2020 |

- Conners, C. K., Erhardt, D., & Sparrow, E. P. (1999). Conners' adult ADHD rating scales (CAARS): technical manual. North Tonawanda, NY: Multi-Health Systems.
- Nilsson, M. E., Suryawanshi, S., Gassmann-Mayer, C., Dubrava, S., McSorley, P., & Jiang, K. (2013). Columbia–suicide severity rating scale scoring and data analysis guide. CSSRS Scoring Version, 2, 1-13.

## 13. Appendix

13.1 Normal Range of Laboratory Tests

Clinical Laboratories, Department of Laboratory Medicine, the Medical Center at the University of California, San Francisco, CA 94143.

- 2019-08-15
- 2020-02-01
- 13.2 Mock-up Tables
- 13.3 Mock-up Patient Data Listings